CLINICAL TRIAL: NCT06933745
Title: Ultrasound of Carotid and Femoral Plaque Burden and Non-alcoholic Fatty Liver Disease as Predictors of Cardiovascular Disease
Brief Title: Ultrasound Assessment of Atherosclerotic Plaque Burden and Cardiovascular Risk: A 10-Year Prospective Study
Acronym: P-SONAR
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Jonn Terje Geitung, Professor, University of Oslo
Other Study IDs: Ahus, BDA
Record Dates: First submitted 2025-04-08; First posted 2025-04-18 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases; Fatty Liver; Atherosclerosis of Femoral Artery; Carotid Artery Plaque; Stroke; Ischemic Cardiovascular Disease; Atheroscleroses
Keywords: Ultrasound; Carotid arteries; Femoral arteries; Cardiovascular Disseases; Plaque burden; Subclinical atherosclerosis; NORRISK2; Ischemic stroke; Ischemic heart disease; Atherosclerotic cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases; Fatty Liver; Carotid Stenosis; Stroke; Atherosclerosis; Ischemic Stroke; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants undergoing ultrasound and screening for conventional CV risk factors.: A sub-cohort consists of 5 500 participants who undergo both carotid and femoral ultrasound and fatty liver status assessment by ultrasound, in addition to assessement of traditional CV risk factors including history of smoking, total-cholesterol, LDL-cholesterol, HDL-cholesterol, Lp(a), blood glucose, systolic and diastolic blood pressure and waist circumference measurements.
- Participants undergoing ultrasound examination: Total cohort consists of 22 000 participants who undergo both carotid and femoral ultrasound and fatty liver status assessment by ultrasound

SUMMARY:
The P-SONAR study is a large, observational, prospective cohort study. The overall aim of the study is to investigate whether plaque burden estimation by 2D ultrasound of the carotid and femoral arteries may enhance cardiovascular risk prediction beyond NORRISK-2

DETAILED DESCRIPTION:
Design: The P-SONAR Study is a prospective cohort study of all men and women aged 45-74 years attending a health check at one of 10 ultrasound clinics in Norway.

Time schedule: Study inclusion and baseline examinations took place in the period April 2022- March 20025.

Current status: Ultrasound follow-up examinations take place from January 2025 - December 2029.

ELIGIBILITY:
Inclusion Criteria: Persons attending a health check during the study period.

-

Exclusion Criteria:

* If they do not consent to participate

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population comprises consecutive persons 45-74 years self-reffered for a health check in one of 10 ultrasound clinics in Norway.
Sampling Method: Non-Probability Sample
Enrollment: 21029 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Carotid and femoral plaque burden cardiovascular (CV) predictive ability beyond NORRISK-2 | From enrollment to an average of 10 years
  Additative ability of carotid and femoral plaque burden assessed by ultrasound to predict incident cardiovascular events, beyond conventional risk factors by NORRISK-2
May plaque burden predict incident cardiovascular disease. | From enrollment to an average of 10 years.
  Find best cutoff value of wTPT plaque burden to predict incident CV disease, across different age groups and sex.

CONTACTS AND LOCATIONS:
Overall Officials: Jonn-Terje Geitung, MD, PhD, MHA, Principal Investigator — University of Oslo; Serena N.H. Tonstad, MD, PhD, Study Director — Oslo University Hospital
Locations (1):
- Austad Diagnostikk, Oslo, East, Norway

IPD SHARING:
Plan to Share IPD: No
Because of the sensitive nature of the data in this study, participants were assured that raw data would remain confidential and would not be shared.